CLINICAL TRIAL: NCT03648879
Title: Phase II Study Evaluating Confocal Endoscopic Microscopy for Detection of Early Stage Gastric Cancer in Subjects With Hereditary Diffuse Gastric Cancer Syndrome
Brief Title: Confocal Endoscopic Microscopy for Detection of Early Stage Gastric Cancer in Subjects With Hereditary Diffuse Gastric Cancer Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeremy Davis, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 180141; 18-C-0141
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Results first posted 2021-03-25 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Gastric Cancer; Gastric Neoplasms
Keywords: Diagnostic; Diagnosis; EGD; Examination of Stomach
MeSH Terms: conditions — Stomach Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 1/Arm 1 - Upper white-light endoscopy and confocal endoscopic microscopy (Experimental): Upper white-light endoscopy and confocal endoscopic microscopy
  Interventions: Device: Endoscope+Cellvizio(R) 100 microscope

INTERVENTIONS:
Device: Endoscope+Cellvizio(R) 100 microscope — Patients will undergo white-light, upper endoscopy. In addition, during this endoscopy patients will undergo Confocal Endoscopic Microscopy (CEM) using the Cellvizio probe (Mauna Kea Technologies) to scan the same anatomic zones.

SUMMARY:
Background:

People with hereditary gastric cancer syndrome are at increased risk of getting cancer in their stomach. These people should have regular endoscopies and biopsies to check for cancer if they are choosing to keep their stomach. Researchers want to see if they can improve the detection of cancer by endoscopy. Improved endoscopies could better detect early signs of cancer in people with this syndrome.

Objective:

To see if a small microscope attached to an endoscope to inspect the stomach lining is better than regular endoscopy to find the first signs of cancer in the stomach.

Eligibility:

People ages 18 and older who have a personal or family history of a hereditary gastric cancer syndrome or have a mutation that is known to lead to gastric cancer

Design:

Participants will be screened over the phone or in person with:

* Personal and family medical history
* Review of their medical records

Participants will have a physical exam. Then they will be put under general anesthesia. They will have an endoscopy. A lighted tube will be inserted into the mouth and go down to the stomach. First, the standard device will be used. Then participants will be injected with fluorescein. This is a contrast agent. Then the microscope will be added to the tube and the endoscopic evaluation of the stomach will be repeated. During the procedure, biopsies will be taken from different areas of the stomach. Participants will be observed for a few hours after the procedure.

About 14 days after the endoscopy, participants will be asked to return to the clinic for a follow-up visit. This visit can also be conducted over the phone.

DETAILED DESCRIPTION:
Background:

Hereditary Diffuse Gastric Cancer (HDGC) syndrome is caused by a germline mutation in the Cadherin 1 (CDH1) gene. Carriers of this mutation have a 56-70% lifetime risk of developing gastric adenocarcinoma. Current international guidelines recommend endoscopic screening of CDH1 mutation carriers that consists of systematic biopsies of an otherwise normal appearing stomach. However, this approach lacks sufficient sensitivity for detecting intramucosal foci of signet ring cells (SRC), which are pathognomonic of HDGC syndrome. The goal of the current study is to utilize confocal endoscopic microscopy (CEM) for screening the gastric mucosa in this high-risk population.

Objective:

Determine if confocal endoscopic microscopy (CEM) will afford greater sensitivity for detection of signet ring cells (SRC) foci in CDH1 germline mutation carriers.

Eligibility:

CDH1 germline mutation carriers, or those who meet clinical criteria for HDGC testing but have tested negative for a CDH1 gene mutation or those who have other germline mutations suspected to be, or reported to be, associated with HDGC (e.g. Catenin Alpha 1 (CTNNA1).

Design:

Phase II, single-institution study of CEM for detection of intramucosal SRC foci compared to current systematic gastric mapping procedure.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with Cadherin-1 (CDH1) germline mutation known to be pathogenic or likely pathogenic, which may also be classified as "significant" or "likely significant" (patients with variants of "uncertain significance " are excluded)

or

-Patients with Catenin Alpha 1 (CTNNA1) and partner and localizer of breast cancer 2 (BRCA2) (PALB2) germline mutations suspected to be, or reported to be, associated with hereditary diffuse gastric cancer (HDGC) syndrome.

or

* In the absence of a germline CDH1 mutation, patients must meet clinical criteria for genetic testing due to a history suggestive of Hereditary Diffuse Gastric Cancer (HDGC) syndrome
* Age greater than or equal to 18 years.
* Physiologically able to undergo upper endoscopy.
* Ability to understand and the willingness to sign a written informed consent document.
* Pregnant women are eligible during second trimester of pregnancy if clinically indicated for evaluation of cancer.

EXCLUSION CRITERIA:

* Current use of therapeutic anticoagulation medication
* Known bleeding disorder or thrombocytopenia.
* Unstable angina or recent (within 3 months) myocardial infarction
* Any clinical contraindication to general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy L Davis, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the study protocol, statistical analysis plan, and clinical study report.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For 2 years from date of study completion.
Access Criteria: Requests must be made by clinical investigators with interest and/or expertise in gastrointestinal cancers or endoscopic surveillance techniques.

REFERENCES:
- [Result] Schueler SA, Gamble LA, Curtin BF, Ruff SM, Connolly M, Hannah C, Quezado M, Miettinen M, George M, Blakely AM, Hernandez JM, Heller T, Koh C, Davis JL. Evaluation of confocal laser endomicroscopy for detection of occult gastric carcinoma in CDH1 variant carriers. J Gastrointest Oncol. 2021 Apr;12(2):216-225. doi: 10.21037/jgo-20-430. PMID 34012620
- [Derived] Ruff S, Curtin B, Quezado M, Heller T, Koh C, Steinberg SM, Connolly M, Hernandez JM, Davis JL. Evaluation of confocal endoscopic microscopy for detection of early-stage gastric cancer in hereditary diffuse gastric cancer (HDGC) syndrome. J Gastrointest Oncol. 2019 Jun;10(3):407-411. doi: 10.21037/jgo.2019.01.04. PMID 31183189
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0141.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1/Arm 1 - Upper White-light Endoscopy and Confocal Endoscopic Microscopy
Started | 37
Completed | 36
Not Completed | 1
Not completed — Subject determined to have Cadherin-1 (CDH1) variant of uncertain significance. | 1

BASELINE CHARACTERISTICS:
Arm/Group | 1/Arm 1 - Upper White-light Endoscopy and Confocal Endoscopic Microscopy
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.51 (14.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 31
  Ethnicity Unknown or Not Reported | 2
  White | 33
  Race Other | 2
  Race Unknown | 2
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Detectable Confocal Endoscopic Microscopy (CEM) w/Greater Sensitivity for Detection of Signet Ring Cells (SRC)Foci in Cadherin-1 (CDH1) Germline Mutation Carriers Compared to Current Method of Standard White Light Endoscopy
Description: Sensitivity for detection of SRC foci in CDH1 germline mutation carriers was assessed by confocal endoscopic microscopy (CEM) compared to the current method of and standard white light endoscopy.
  Sensitivity in CEM and WLE is defined as the percentage of participants with detectable cancer on endoscopic biopsy.
Time Frame: 14 days
Population: 36/37 were evaluable for this outcome measure. One participant was determined to have Cadherin-1 (CDH1) variant of uncertain significance.
Measure: Number; unit: Percentage of participants
Arm/Group | 1/Arm 1 - Upper White-light Endoscopy and Confocal Endoscopic Microscopy
Number analyzed (Participants) | 36
Percentage of participants
  CEM | 16.7
  White Light Endoscopy | 11.1

2. Secondary Outcome: Percentage of Participants Who Have Signet Ring Cells (SRC) Foci Not Identified by Confocal Endoscopic Microscopy (CEM)
Description: In participants who choose to undergo prophylactic total gastrectomy with permanent pathologic analysis, the false negative rate (the fraction of participants who have SRC foci not identified by CEM and White Light Endoscopy techniques) will be determined and reported. The fraction percentage of patients who underwent prophylactic total gastrectomy with findings of SRC foci in the gastrectomy specimen will represent the denominator (number) and the number of patients with negative findings by CEM and White Light Endoscopy (WLE) will represent the numerator (number) to generate the false negative detection rate (fraction) for CEM and WLE, respectively.
Time Frame: Date of enrollment to date of prophylactic gastrectomy, approximately 6 months or an average of 1 month up to 12 months.
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 1/Arm 1 - Upper White-light Endoscopy and Confocal Endoscopic Microscopy
Number analyzed (Participants) | 36
Percentage of participants
  CEM | 67
  White Light Endoscopy | 87

3. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date of enrollment to date off study, approximately 11 months and 19 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Arm 1 - Upper White-light Endoscopy and Confocal Endoscopic Microscopy
Number analyzed (Participants) | 36
Participants | 1

ADVERSE EVENTS:
Time Frame: Date of enrollment to date off study, approximately 11 months and 19 days.
Description: 36/37 were evaluable for adverse events. One participant was determined to have Cadherin-1 (CDH1) variant of uncertain significance.
Arm/Group | 1/Arm 1 - Upper White-light Endoscopy and Confocal Endoscopic Microscopy
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Arm 1 - Upper White-light Endoscopy and Confocal Endoscopic Microscopy (N=36)
Fever (General disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT03648879/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT03648879/ICF_001.pdf